CLINICAL TRIAL: NCT06187909
Title: Ultrasound-Guided Modified Pectoral Plane (PECS II) Block Versus Midpoint Transverse Process to Pleura (MTP) Block for Postoperative Analgesia of Modified Radical Mastectomy
Brief Title: PECS II vs. MTP for Analgesia After MRM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed abdelghany Khalifa ragab, lecturer of Anesthesia, intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU MD311/2023
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasm Female; Postoperative Pain Management
Keywords: Anesthesia, Conduction; Mastectomy, Modified Radical; Breast Neoplasms; Postoperative Pain; Analgesia, Opioid; Nerve Block
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment model involving 88 ASA I-II female patients undergoing modified radical mastectomy. Participants were randomized into two equal groups to receive either an ultrasound-guided PECS II block or a midpoint transverse process to pleura (MTP) block, each with 20 mL of 0.25% bupivacaine. Postoperative analgesic efficacy was assessed using the Visual Analog Scale (VAS), time to first rescue analgesia, total nalbuphine consumption, and incidence of complications over 24 hours.
Who Masked: Outcomes Assessor
Masking Description: Patients were sedated during block placement; however, due to the distinct anatomical sites of the two techniques, full patient blinding could not be ensured. Outcome assessors gathering postoperative data were blinded to group allocation, and the anesthesiologists performing the blocks were not engaged in data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PECS II block group (Active Comparator): Forty-four female patients (ASA I-II, 40-65 years) scheduled for modified radical mastectomy received an ultrasound-guided PECS II block with 20 mL of 0.25% bupivacaine (10 mL between pectoralis major and minor; 10 mL between pectoralis minor and serratus anterior).
  Interventions: Procedure: PECS II BLOCK
- MTP block group (Active Comparator): Forty-four female patients (ASA I-II, 40-65 years) scheduled for modified radical mastectomy received an ultrasound-guided midpoint transverse process to pleura (MTP) block with 20 mL of 0.25% bupivacaine (10 mL injected at T2 and 10 mL at T6).
  Interventions: Procedure: MTP BLOCK

INTERVENTIONS:
Procedure: PECS II BLOCK — In the supine position, as described by Blanco et al., the ultrasound probe was placed transversely beneath the clavicle. After identifying the intermuscular plane between the pectoralis major and minor, 10 mL of 0.25% bupivacaine was injected. The probe was then repositioned laterally to identify the plane between the pectoralis minor and serratus anterior at the third to fourth ribs, where a further 10 mL of 0.25% bupivacaine was injected.
  Arms: PECS II block group
Procedure: MTP BLOCK — The block was performed with the patient in a seated position. The ultrasound probe was positioned parasagittally, approximately 3 cm lateral to the midline, at the T2 and T6 vertebral levels. A 22-gauge needle was advanced in-plane to the midpoint between the transverse process and pleura, and 10 mL of 0.25% bupivacaine was injected at each level. This protocol was adapted from the original technique described by Bhoi et al., with modifications in injection levels and volume.
  Arms: MTP block group

SUMMARY:
This randomized controlled study aims to compare the analgesic efficacy of the ultrasound-guided modified pectoral nerve block (PECS II) and the midpoint transverse process to pleura (MTP) block in female patients undergoing modified radical mastectomy (MRM). Postoperative pain intensity will be assessed using the Visual Analog Scale (VAS) over the first 24 hours, with additional evaluation of opioid consumption and complications.

DETAILED DESCRIPTION:
Modified radical mastectomy (MRM) is associated with significant postoperative pain, which may increase opioid use, delay recovery, and contribute to chronic post-mastectomy pain syndrome. This study compares two regional analgesic techniques: the ultrasound-guided modified pectoral nerve block (PECS II) and the midpoint transverse process to pleura (MTP) block.

The PECS II block involves the injection of local anesthetic between the pectoralis minor and serratus anterior muscles, targeting the pectoral nerves and lateral cutaneous branches of intercostal nerves (T2-T6). It is widely used for anterior chest wall analgesia after breast surgery. The MTP block, a more recent paravertebral-domain technique, deposits anesthetic midway between the transverse process and the pleura, allowing spread to dorsal and ventral rami via the superior costotransverse ligament and potentially achieving broader thoracic segment coverage.

This randomized trial evaluates postoperative pain control using the Visual Analog Scale (VAS) over 24 hours, along with opioid consumption and adverse events. The aim is to determine whether the MTP block offers superior analgesia and an opioid-sparing effect compared to the PECS II block.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients scheduled for modified radical mastectomy (MRM).
2. Age between 40 and 65 years.
3. American Society of Anesthesiologists (ASA) physical status I-II.

Exclusion Criteria:

1. Known allergy to local anesthetics.
2. Coagulopathy.
3. Infection at the site of injection.
4. Patient refusal.
5. Inability to understand or use the pain scale.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study population restricted to female patients undergoing modified radical mastectomy.
Enrollment: 88 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A. Khalifa, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of institutional policy and patient confidentiality concerns. Only summarized results will be made available in the published manuscript and upon reasonable request.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-center, prospective, randomized controlled trial conducted at Ain Shams University Hospital. A total of 112 patients scheduled for modified radical mastectomy were assessed for eligibility between November 2023 and July 2025.
Pre-assignment Details: Out of 112 screened patients, 24 were excluded (17 did not meet inclusion criteria, 7 declined participation), leaving 88 enrolled and randomly allocated to Group A (PECS II block, n=44) and Group B (MTP block, n=44).
  Four participants withdrew consent during follow-up, resulting in 84 completions (42 per group). All remaining participants were included in the final analysis, with no exclusions
Groups:
- MTP Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy, received an ultrasound-guided midpoint transverse process to pleura (MTP) block. A high-frequency linear probe was placed parasagittally, approximately 3 cm lateral to the midline at the T2 and T6 vertebral levels. A 22-gauge echogenic needle was advanced in-plane to the midpoint between the transverse process and pleura, and 10 mL of 0.25% bupivacaine was injected at each level.
- PECS II Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy, received an ultrasound-guided PECS II block. A high-frequency linear probe was placed beneath the clavicle to identify the intermuscular plane between the pectoralis major and minor, where 10 mL of 0.25% bupivacaine was injected. The probe was then repositioned laterally to identify the plane between the pectoralis minor and serratus anterior at the level of the third to fourth ribs, where another 10 mL of 0.25% bupivacaine was injected.
Period: Overall Study
Arm/Group | MTP Block Group | PECS II Block Group
Started | 44 | 44
Completed | 42 | 42
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- MTP Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy, received an ultrasound-guided midpoint transverse process to pleura (MTP) block. A high-frequency linear probe was positioned parasagittally about 3 cm lateral to the midline at the T2 and T6 vertebral levels. A 22-gauge needle was advanced in-plane, and 10 mL of 0.25% bupivacaine was injected at each level.
- PECS II Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy, received an ultrasound-guided PECS II block with 20 mL of 0.25% bupivacaine (10 mL between the pectoralis major and minor, and 10 mL between the pectoralis minor and serratus anterior at the third to fourth ribs).
- Total: Total of all reporting groups
Arm/Group | MTP Block Group | PECS II Block Group | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (5.8) | 41.2 (4.9) | 41.8 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 42 | 84
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
weight [Mean (Standard Deviation); unit: kilograms] | 78.5 (8.5) | 79.1 (8.5) | 78.8 (8.5)
height [Mean (Standard Deviation); unit: meters] | 1.68 (0.06) | 1.67 (0.05) | 1.675 (0.055)
body mass index [Mean (Standard Deviation); unit: kilograms per meter square] | 27.9 (2.3) | 28.3 (2.2) | 28.1 (2.25)

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Pain Severity Assessed by VAS at Hour-4
Description: Visual Analogue Scale is a scale for pain assessment ranging from 0 to 10 where 0 is minimum and means no pain while 10 is maximum and means maximum pain which means worse outcome
Time Frame: will be evaluated at hour-4 postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- MTP Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy received an ultrasound-guided midpoint transverse process to pleura (MTP) block. A high-frequency linear probe was positioned parasagittally about 3 cm lateral to the midline at the T2 and T6 vertebral levels. A 22-gauge echogenic needle was advanced in-plane to the midpoint between the transverse process and pleura, and 10 mL of 0.25% bupivacaine was injected at each level.
- PECS II Block Group: Forty-four ASA I-II female patients, aged 40-65 years and scheduled for modified radical mastectomy, received an ultrasound-guided PECS II block. Using a high-frequency linear probe, 10 mL of 0.25% bupivacaine was injected between the pectoralis major and minor muscles. The probe was then repositioned laterally to the plane between the pectoralis minor and serratus anterior at the third to fourth ribs, where another 10 mL of 0.25% bupivacaine was injected.
Arm/Group | MTP Block Group | PECS II Block Group
Number analyzed (Participants) | 42 | 42
score on a scale | 1.4 (0.6) | 2.2 (0.7)

2. Secondary Outcome: Post-operative Pain Severity Assessed by VAS on Admission to Postanesthesia Care Unit (PACU), at Hour-2, Hour-8, Hour-12, Hour-18 and Hour-24.
Description: Comparison between postoperative pain severity after 2 hours, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours postoperative between both groups using visual analogue score Visual Analogue Scale is a scale for pain assessment ranging from 0 to 10 where 0 is minimum and means no pain while 10 is maximum and means maximum pain which means worse outcome
Time Frame: 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MTP Block Group | PECS II Block Group
Number analyzed (Participants) | 42 | 42
score on a scale
  Post-operative pain severity assessed by Visual analogue scale on admission to PACU | 0.3 (0.5) | 0.3 (0.5)
  Post-operative pain severity assessed by Visual analogue scale at 2 hours postoperatively. | 1.1 (0.8) | 1.4 (0.6)
  Post-operative pain severity assessed by Visual analogue scale at 8 hours postoperatively. | 2.5 (0.5) | 3.2 (0.6)
  Post-operative pain severity assessed by Visual analogue scale at 12 hours postoperatively. | 2.9 (0.6) | 3.2 (0.7)
  Post-operative pain severity assessed by Visual analogue scale at 18 hours postoperatively. | 1.9 (0.7) | 2.2 (0.5)
  Post-operative pain severity assessed by Visual analogue scale at 24 hours postoperatively. | 1.5 (0.8) | 1.7 (0.5)

3. Secondary Outcome: Time of First Rescue Analgesia
Description: Comparison between both groups regarding the time of first needed dose of nalbuphine
Time Frame: 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | MTP Block Group | PECS II Block Group
Number analyzed (Participants) | 42 | 42
hours | 12.8 (0.8) | 7.9 (1.2)

4. Secondary Outcome: Cumulative Post-operative Nalbuphine Consumption in the First 24 Hours
Description: Comparison between both groups regarding total consumed nalbuphine in first 24 hours postoperative
Time Frame: 24 hours postoperatively
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | MTP Block Group | PECS II Block Group
Number analyzed (Participants) | 42 | 42
milligrams | 8.3 (2.6) | 13.3 (3.6)

5. Secondary Outcome: Incidence of Postoperative Side Effects and Complications
Description: Comparison between both groups regarding postoperative side effects and complications
Time Frame: 24 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | MTP Block Group | PECS II Block Group
Number analyzed (Participants) | 42 | 42
Participants
  Hematoma | 9 | 12
  Nausea | 2 | 8
  vomiting | 1 | 3
  pneumothorax | 1 | 0

ADVERSE EVENTS:
Time Frame: 24 hours postoperatively
Description: Adverse events included block-related complications: vascular puncture, pneumothorax, and local anesthetic systemic toxicity. Events were assessed by anesthesiologists intraoperatively and during the first 24 hours after surgery.
Arm/Group | MTP Block Group | PECS II Block Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42 | 0/42
Other Adverse Events (participants affected / at risk) | 12/42 | 23/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTP Block Group (N=42) | PECS II Block Group (N=42)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTP Block Group (N=42) | PECS II Block Group (N=42)
Hematoma (Injury, poisoning and procedural complications) | 9 (9) | 12 (12)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT06187909/Prot_SAP_002.pdf